CLINICAL TRIAL: NCT00569114
Title: A Phase 1 Dose-Escalation Pharmacokinetic and Pharmacodynamic Study of TG01 Tablets in Combination With Erlotinib in Non-Small Cell Lung Cancer Patients
Brief Title: Phase 1 Study of TG01 and Erlotinib in Non-small Cell Lung Cancer (NCSLC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sara Zaknoen, MD, Tragara Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TP2001-101
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: TG01

INTERVENTIONS:
Drug: TG01 — Drug:TG01tablets given orally QD Drug: erlotinib tablets 150mg QD

SUMMARY:
This is a multicenter, open-label, phase 1, dose escalation study. The purpose is to determine the highest dose of TG01 that can be safely given to patients with Non-Small Cell Lung Cancer in combination with erlotinib.

ELIGIBILITY:
Inclusion Criteria (include but are not limited to):

* Histogically or pathologically determined relapsed/recurrent Stage IIIb (plueral effusion) or IV NSCLC.
* Measurable or evaluable disease as defined by RECIST
* Must have failed at least one prior chemotherapy regimen or have refused chemotherapy.
* ECOG perfromance status of 0,1, or 2.

Exclusion Criteria (include but are not limited to):

* Radiation therapy (excluding CNS therapy) < 2 weeks, chemotherapy, non-cytotoxic investigational agents or high dose corticosteroids within 3 weeks of intitating therpy or patients who have not recovered from adverse effects due to agents administered more than 3 weeks earlier.
* Evidence of New York Heart Associatation Class III or greater cardiac disease.
* History of myocardial infarction, stroke, or cardiovascular intervention within the last 12 months.
* Patients on anti-platlet drugs or anticoagulants such as Placix and Coumadin.
* Systemic central nervous system metastases. The patient must be stable after radiotherapy for >/= to 2 weeks and off corticosteroids for >/= to 1 week.
* Pregnant or nursing women.
* Patients who are primarily refactory to erlotinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Saftey, maximum tolerated dose, optimal biological dose and pharmacokinetics. | Baseline, 8, 15 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara Zaknoen, MD, Study Director — Tragara Pharmaceuticals
Locations (5):
- United States (5):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - University of California at Davis, Sacramento, California
  - Nevada Cancer Institute, Las Vegas, Nevada